CLINICAL TRIAL: NCT03337087
Title: Phase I Study of Irinotecan Liposome (Nal-IRI), Fluorouracil and Rucaparib in the Treatment of Select Gastrointestinal Metastatic Malignancies Followed by a Phase Ib of First and Second Line Treatment of Both Unselected and Selected (for BRCA 1/2 and PALB2 Mutations) Patients With Metastatic Adenocarcinoma of the Pancreas Then Followed by a Phase II Study of First Line Treatment of Selected Patients With Metastatic Adenocarcinoma of the Pancreas With Genomic Markers (Signature) of Homologous Recombination Deficiency (HRD)
Brief Title: Liposomal Irinotecan, Fluorouracil, Leucovorin Calcium, and Rucaparib in Treating Patients With Metastatic Pancreatic, Colorectal, Gastroesophageal, or Biliary Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-GI-1603; NCI-2017-01976 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-GI-1603 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Metastatic Biliary Tract Carcinoma; Metastatic Colorectal Carcinoma; Metastatic Gastroesophageal Junction Adenocarcinoma; Metastatic Malignant Digestive System Neoplasm; Metastatic Pancreatic Adenocarcinoma; Stage IV Colorectal Cancer AJCC v7; Stage IV Pancreatic Cancer AJCC v6 and v7; Stage IVA Colorectal Cancer AJCC v7; Stage IVB Colorectal Cancer AJCC v7
MeSH Terms: conditions — Colorectal Neoplasms; Gastrointestinal Neoplasms | interventions — Fluorouracil; dehydroftorafur; irinotecan sucrosofate; Leucovorin; rucaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (nal-IRI, leucovorin, fluorouracil, rucaparib) (Experimental): PHASE Ia: Patients receive liposomal irinotecan IV over 90 minutes, leucovorin calcium IV, and fluorouracil IV over 46 hours on days 1 and 15. Patients also receive rucaparib PO BID on days 4-13 and 18-27. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity.
  PHASE Ib/II: Patients receive liposomal irinotecan IV over 90 minutes and fluorouracil IV over 46 hours on days 1 and 15. Patients also receive rucaparib PO BID on days 4-13 and 18-27. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity.
  Interventions: Drug: Fluorouracil; Drug: Irinotecan Sucrosofate; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Rucaparib

INTERVENTIONS:
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Irinotecan Sucrosofate — Given IV
  Other Names: Irinotecan Liposome; MM-398; nal-IRI; Nanoliposomal Irinotecan; Nanoparticle Liposome Formulation of Irinotecan; Onivyde; PEP02
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Rucaparib — Given PO
  Other Names: 6H-Pyrrolo(4,3,2-ef)(2)benzazepin-6-one, 8-Fluoro-1,3,4,5-tetrahydro-2-(4-((methylamino)methyl)phenyl)-; 8-Fluoro-2-(4-((methylamino)methyl)phenyl)-1,3,4,5-tetrahydro-6H-azepino(5,4,3-cd)indol-6-one

SUMMARY:
This phase I/II trial studies the side effects and best dose of liposomal irinotecan and rucaparib when given together with fluorouracil and leucovorin calcium and to see how well they work in treating patients with pancreatic, colorectal, gastroesophageal, or biliary cancer that has spread to other places in the body (metastatic). Chemotherapy drugs, such as liposomal irinotecan, fluorouracil, and leucovorin calcium, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. PARPs are proteins that help repair DNA mutations. PARP inhibitors, such as rucaparib, can keep PARP from working, so tumor cells can't repair themselves, and they may stop growing. Giving liposomal irinotecan and rucaparib together with fluorouracil and leucovorin calcium may work better in treating patients with pancreatic, colorectal, gastroesophageal, or biliary cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the recommended dose level for the phase Ib and phase II trial of liposomal irinotecan (nal-IRI) and fluorouracil (5-FU) with rucaparib (MFR) in patients with metastatic disease from pancreatic cancer (up to 2 lines of prior therapy), colorectal cancer (up to 3 lines of prior therapy), gastroesophageal cancer (up to 1 line of prior therapy) and biliary tract cancer (with 1 line of prior therapy allowed). (Phase I) II. To assess, in a preliminary fashion, antitumor efficacy, in terms of disease control rate and further tolerability, of the recommended dose level of combination of nal-IRI and 5-FU with rucaparib in patients with metastatic disease from pancreatic cancer (=< 1 line of prior therapy in the metastatic setting). (Phase Ib) III. To estimate the proportion of evaluable patients who reach complete response (CR)/partial response (PR) =< 32 weeks after registration among patients with metastatic adenocarcinoma of the pancreas with genomic markers (signature) of homologous recombination deficiency (HRD), specifically BRCA1, BRCA2, and PALB2 mutation, treated with the combination of nal-IRI and 5FU with rucaparib (MFR). (Phase II)

SECONDARY OBJECTIVES:

I. To estimate the progression-free survival (PFS) and overall survival (OS) for patients with metastatic adenocarcinoma of the pancreas with genomic markers (signature) of homologous recombination deficiency (HRD), specifically BRCA1, BRCA2, and PALB2 mutation, treated with the combination of nal-IRI and 5-FU with rucaparib (MFR). (Phase II) II. To assess the toxicity of the combination of nal-IRI and 5-FU with rucaparib in patients with metastatic adenocarcinoma of the pancreas with genomic markers (signature) of homologous recombination deficiency (HRD), specifically BRCA1/2 and PALB2 mutations. (Phase II)

EXPLORATORY OBJECTIVES:

I. To evaluate the role of genomic markers (signature) of HRD, mutation other than BRCA1, BRCA2, and PALB2 as predictive biomarkers of response to MFR.

II. To evaluate BRCA1, BRCA2, and PALB2 mutations as predictive biomarker of response to MFR.

OUTLINE: This is phase I, dose-escalation study of liposomal irinotecan and rucaparib and followed by a phase II study.

PHASE Ia: Patients receive liposomal irinotecan intravenously (IV) over 90 minutes, leucovorin calcium IV, and fluorouracil IV over 46 hours on days 1 and 15. Patients also receive rucaparib orally (PO) twice daily (BID) on days 4-13 and 18-27. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity.

PHASE Ib/II: Patients receive liposomal irinotecan IV over 90 minutes and fluorouracil IV over 46 hours on days 1 and 15. Patients also receive rucaparib PO BID on days 4-13 and 18-27. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity.

After completion of study treatment, patients are followed up every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Phase I only: Histologic confirmation of pancreatic, colorectal, gastroesophageal or biliary adenocarcinoma, as follows:

  * Patients with metastatic disease from pancreatic cancer who received no more than 2 lines of prior therapy in the metastatic setting
  * Patients with metastatic disease from colorectal cancer who received no more than 3 lines of prior therapy in the metastatic setting
  * Patients with metastatic disease from gastroesophageal cancer who received no more than 1 line of prior therapy in the metastatic setting
  * Patients with metastatic disease from biliary tract cancer who received no more than 1 line of prior therapy in the metastatic setting
  * NOTE: No prior exposure to irinotecan in the metastatic setting will be allowed except in the phase I dose escalation portion and in colon cancer patients only; in pancreas cancer, exposure to irinotecan is only allowed in the neoadjuvant setting and no progressive disease < 3 months from last dose of irinotecan
* Phase Ib only: Patients with metastatic adenocarcinoma of the pancreas who have who received no more than 1 line of prior therapy in the metastatic setting

  * NOTE: Exposure to irinotecan is only allowed in the neoadjuvant setting and no progressive disease < 3 months from last dose of irinotecan
* Phase II only: Patients with metastatic adenocarcinoma of the pancreas with genomic markers (signature) of homologous recombination deficiency (HRD) or BRCA1 or BRCA2 or PALB2 mutation, or HRD (non-BRCA, non-PALB) who have not received any systemic therapy in the metastatic setting

  * NOTE: Exposure to irinotecan is only allowed in the neoadjuvant setting and no progressive disease < 3 months from last dose of irinotecan
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 21 days prior to registration)
* Platelet count >= 100,000/mm^3 (obtained =< 21 days prior to registration)
* Hemoglobin > 9.0 g/dL (obtained =< 21 days prior to registration)
* Total bilirubin =< institutional upper limit of normal (ULN) (obtained =< 21 days prior to registration)
* Aspartate transaminase (AST) =< 3 x ULN, =< 5.0 x ULN for patients with metastatic disease to the liver (obtained =< 21 days prior to registration)
* Aminotransferase (ALT) =< 3.0 x ULN, =< 5.0 x ULN for patients with metastatic disease to the liver (obtained =< 21 days prior to registration)
* Creatinine =< 1.0 mg/dL or creatinine clearance >= 45 ml/min using the Cockcroft-Gault formula (obtained =< 21 days prior to registration)
* Negative serum or urine pregnancy test done =< 7 days prior to registration and repeated prior to dosing on day 1 of each cycle, for individuals of childbearing potential only; NOTE: Individuals are considered to be of childbearing potential unless one of the following applies:

  * Is postmenopausal, defined as no menses for at least 12 months without an alternative medical cause; a high follicle-stimulating hormone (FSH) level consistently in the postmenopausal range (30 mIU/mL or higher) may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy; however, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient to confirm a postmenopausal state: or
  * Considered to be permanently sterile; permanent sterilization includes hysterectomy, bilateral salpingectomy, and/or bilateral oophorectomy
* Provide informed written consent
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)

  * Note: During the active monitoring phase of a study (i.e., active treatment and observation), participants must be willing to return to the consenting institution for follow-up
* Willing to provide tissue and blood samples for mandatory correlative research purposes
* Individuals of reproductive potential and their partners willing to practice total abstinence or use a highly effective method of contraception (failure rate < 1% per year) during treatment and for 6 months following the last dose of rucaparib; the following are allowable only:

  * Ongoing use of progesterone-only injectable or implantable contraceptives (eg, Depo Provera, Implanon, Nexplanon)
  * Placement of an intrauterine device or intrauterine system
  * Bilateral tubal occlusion
  * Sterilization, with appropriate post-vasectomy documentation of absence of sperm in ejaculate
  * True, complete (as opposed to periodic) abstinence
* Patients must discontinue prior chemotherapy >= 28 days before registration

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant individuals
  * Nursing individuals
  * Persons of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Previous or concurrent cancer that is distinct in primary site or histology from cancer of primary site =< 3 years prior to registration EXCEPT for curatively treated cervical cancer in situ, melanoma in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)]; Note: All cancer treatments for those distinct in a primary site other than cancer of origin must be completed >= 3 years prior to registration
* Received any prior poly ADP-ribose polymerase inhibitor (PARPi) treatment. Patients who received prior PARPi treatment in the adjuvant setting with the last dose received more than 12 months prior to registration are allowed to enroll.
* Corrected QT interval (QTc) prolongation > 480 msec, as calculated by either the Bazett or Fridericia formula, as per institutional standard
* Inability to swallow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2025-08-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tanios S Bekaii-Saab, Principal Investigator — Academic and Community Cancer Research United
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Mayo Clinic in Rochester, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Nal-IRI, Leucovorin, Fluorouracil, Rucaparib): PHASE Ia: Patients receive liposomal irinotecan IV over 90 minutes, leucovorin calcium IV, and fluorouracil IV over 46 hours on days 1 and 15. Patients also receive rucaparib PO BID on days 4-13 and 18-27. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity.> > PHASE Ib/II: Patients receive liposomal irinotecan IV over 90 minutes and fluorouracil IV over 46 hours on days 1 and 15. Patients also receive rucaparib PO BID on days 4-13 and 18-27. Cycles repeat every 28 days in the absence of disease progression or unaccepted toxicity.>
  > Fluorouracil: Given IV>
  > Irinotecan Sucrosofate: Given IV>
  > Laboratory Biomarker Analysis: Correlative studies>
  > Leucovorin Calcium: Given IV>
  > Rucaparib: Given PO
Period: Overall Study
Arm/Group | Treatment (Nal-IRI, Leucovorin, Fluorouracil, Rucaparib)
Started | 18
Completed | 12
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nal-IRI, Leucovorin, Fluorouracil, Rucaparib)
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 55.0 [35.0 to 70.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  All Other | 1
  White | 17
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG = 0: Fully active, able to carry on all pre-disease performance without restriction. > ECOG = 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. > ECOG = 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours. > ECOG = 0 is better. ECOG = 2 is worse.
  Participants
    0 | 6
    1 | 12
Histologic grade (differentiation) [Count of Participants; unit: Participants]
  G1 (Well differentiated) | 1
  G2 (Moderately differentiated) | 9
  G3 (Poorly differentiated) | 2
  GX (Grade cannot be assessed) | 6
Number of Metastatic Sites [Count of Participants; unit: Participants]
  1 | 6
  2 | 6
  3+ | 6
Cancer Type [Count of Participants; unit: Participants]
  Colorectal | 11
  Gastroesophageal | 1
  Pancreatic | 6
Prior Systemic Therapies in Metastatic Setting [Count of Participants; unit: Participants]
  0 | 5
  1 | 2
  2 | 7
  3 | 3
  4+ | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (Phase I)
Description: Will be assessed to determine maximum tolerated dose (MTD) of the combination of liposomal irinotecan (nal-IRI) and fluorouracil (5FU) with rucaparib (MFR). MTD is defined as the dose level below the lowest dose that induces dose-limiting toxicity (DLT) in at least one-third of patients (at least 2 of a maximum of 6 new patients). A total of 6 patients treated at the MTD will be sufficient to identify common toxicities at the MTD.
Time Frame: Up to 28 days from start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nal-IRI, Leucovorin, Fluorouracil, Rucaparib)
Number analyzed (Participants) | 12
Participants | 1

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Treatment (Nal-IRI, Leucovorin, Fluorouracil, Rucaparib)
All-Cause Mortality (participants affected / at risk) | 1/18
Serious Adverse Events (participants affected / at risk) | 15/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nal-IRI, Leucovorin, Fluorouracil, Rucaparib) (N=18)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (6)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (4)
Obstruction gastric (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (3)
Fever (General disorders) | 3 (4)
Multi-organ failure (General disorders) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (3)
Neutrophil count decreased (Investigations) | 4 (4)
Platelet count decreased (Investigations) | 1 (2)
White blood cell decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nal-IRI, Leucovorin, Fluorouracil, Rucaparib) (N=18)
Anemia (Blood and lymphatic system disorders) | 12 (51)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Periorbital edema (Eye disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 13 (66)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 2 (6)
Gastrointestinal fistula (Gastrointestinal disorders) | 1 (3)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 13 (55)
Oral pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (20)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 6 (8)
Fatigue (General disorders) | 12 (91)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (2)
Alanine aminotransferase increased (Investigations) | 8 (24)
Alkaline phosphatase increased (Investigations) | 15 (65)
Aspartate aminotransferase increased (Investigations) | 8 (23)
Blood bilirubin increased (Investigations) | 5 (11)
Creatinine increased (Investigations) | 4 (7)
Lymphocyte count decreased (Investigations) | 8 (50)
Neutrophil count decreased (Investigations) | 11 (23)
Platelet count decreased (Investigations) | 9 (31)
Weight loss (Investigations) | 3 (3)
White blood cell decreased (Investigations) | 11 (17)
Anorexia (Metabolism and nutrition disorders) | 4 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (9)
Hypokalemia (Metabolism and nutrition disorders) | 12 (27)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (5)
Headache (Nervous system disorders) | 3 (5)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (14)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/87/NCT03337087/Prot_SAP_000.pdf